CLINICAL TRIAL: NCT05875064
Title: Aesthetic Restorations in Deciduous Anterior Teeth - Study Protocol for a Randomized Clinical Trial
Brief Title: Aesthetic Restorations in Deciduous Anterior Teeth
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RehabAnteriorUnimes
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — Composite Resins

STUDY DESIGN:
Intervention Model Description: This is a non-inferiority randomized clinical trial with parallel arms, with an allocation ratio of 1:1
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional restoration group (control) (Active Comparator): The teeth allocated in the conventional restoration group (control) will receive restorations in resin composed by incremental technique, using opaque resin. For this, 37% phosphoric acid (Condac37, FGM) will be applied for 15 seconds, and then, after washing and relative drying of the surface, application of universal adhesive (Universal Beautibond Adhesive, Shofu) with the aid of microbrush on the entire dental surface, photoactivation of the adhesive and restoration by incremental technique and photoactivation of each layer of resin for 20 seconds. The tooth will receive finishing and polishing through rotating instruments and abrasive discs (Supersnap, Shofu).
  Interventions: Procedure: Restoration with conventional resin composite
- polyvinyl crown - experimental group (Experimental): The teeth allocated in the experimental group will have the restorations carried out through monochromatic composite resin with chameleon effect in single insertion through polyvinyl crown. For this, 37% phosphoric acid (Condac37, FGM) will be applied for 15 seconds, and then, after washing and relative drying of the surface, application of universal adhesive (Universal Beautibond Adhesive, Shofu) with the aid of microbrush on the entire tooth surface, photoactivation of the adhesive and adaptation of the crown matrix in acetate filled with resin in the tooth. Photoactivation will be done for 20 seconds per dental face, and the acetate matrix is then removed. The tooth will receive finishing and polishing through rotating instruments and abrasive discs (Supersnap, Shofu).
  Interventions: Combination Product: Restoration with resin composite and polyvinyl crown

INTERVENTIONS:
Combination Product: Restoration with resin composite and polyvinyl crown — Restorative treatment of anterior primary teeth with monochromatic composite resin in single insertion through polyvinyl crowns, after selective removal of carious tissue compared to the effectiveness of conventional restoration.
  Arms: polyvinyl crown - experimental group
Procedure: Restoration with conventional resin composite — Restorative treatment of anterior primary teeth with conventional composite resin, after selective removal of carious tissue
  Arms: conventional restoration group (control)

SUMMARY:
This study proposes to conduct a randomized clinical trial (RCT), composed of a sample of 194 deciduous central and lateral incisors with active cavitated lesions, simplified ICDAS C+ score, with involvement of more than two surfaces. This sample will be divided into two experimental groups, both with selective removal of carious tissue: a group in which conventional restoration will be performed using opaque resins; and another group with monochromatic resin with chameleon effect and polyvinyl crowns.

ELIGIBILITY:
Inclusion Criteria:

* Children ranging in age from 12 to 60 months with at least one active cavitated caries lesion involving more than 2 surfaces (C+ score) in deciduous upper incisors will be included.

Exclusion Criteria:

* Patients with special needs, with general health conditions that may affect the oral cavity, whose guardians do not sign the Inform Consent Form will be excluded. In addition, teeth with pulp exposure, spontaneous pain, mobility, presence of swelling or fistula near the tooth and teeth with previous restorations; less than 2/3 of root (radiographically assessed), teeth without an antagonist, teeth with previous restorations and children with bruxism and/or deep bite.

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2025-01-26 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in progression of caries lesion through clinical criteria and longevity of restorations | Baseline and after 6, 12, 18 and 24 months.
  The integrity of the restoration, its adaptation in all dental faces and identified possible failures related to structural fracture, resin wear, maladaptation or functional maintenance of the restored tooth will be verified.
  The clinical evaluation of the retention of the restorations will be performed after 6, 12, 18 and 24 months, using the criteria: total retention; Partial retention 1 - presence of the resin in two thirds of the surface of each dental face; Partial retention 2 - presence of the resin in one third d and each face of the dental surface, total loss of resin on the surface of the dental surface.
  It will also be evaluated the degree of tooth mobility and its relationship with the usual exfoliation period in the teeth belonging to both groups. In teeth where the restoration is intact and clinical features of associated lesions are not verified, the lesions will be considered as inactive.

SECONDARY OUTCOMES:
Change in the progression of caries lesion by radiographic criteria | Baseline and after 6, 12, 18 and 24 months.
  For the evaluation of caries progression, the modified periapical radiographic examination for preschoolers will be used. The images will be compared two by two in order to evaluate whether or not there was progression of caries:
  1. Absent progression: when there is no increase in the radiolucent area of the lesion.
  2. Progression present: when there is an increase in the radiolucent area of the lesion.
  Teeth that present progression of caries lesion to signs of pulp involvement, will receive restorative or endodontic treatment compatible with the observed picture.
Change in the perception of parents/guardians | Baseline and after 6, 12, 18 and 24 months.
  To evaluate the perception of parents/guardians in relation to the treatment performed, the questionnaire "Child's and parent's questionnaire about teeth appearance" will be used soon after the first treatment session and 6 months after the treatment. The examiners will guide you to express your real opinion.
Change in the satisfaction of parents/guardians | Baseline and after 6, 12, 18 and 24 months.
  The parents/guardians will be asked about their satisfaction with the treatment performed on the child. They will answer 5 "yes" or "no" questions about how much they liked the procedures. The examiners will guide you to issue your real opinion after 6 months of treatment.
Change in the impact of treatments on children's oral health-related quality of life | Baseline and after 6, 12, 18 and 24 months.
  A questionnaire will be applied to assess the impact of treatments on children's oral health-related quality of life. The validated Brazilian version of the Early Childhood Oral Health Impact Scale (ECOHIS) should be answered by the parents or guardians of the participants in the initial consultations and at each return. The higher the score, the worse is the children's oral health-related quality of life.

IPD SHARING:
Plan to Share IPD: Yes
Data generated from this clinical trial will be made available to other researchers upon reasonable request. The data will be shared in accordance with BMJ's Tier 2 data policy, ensuring legal and ethical considerations are upheld.
  * Description of Data: The dataset includes anonymized patient records, clinical outcome measures, and intervention details.
  * Availability: Data will be accessible within 6 months of publication of the final study results.
  * Access: Requests for data access can be submitted through OSF.
  * Protection: Personal identifiers will be removed to protect participant confidentiality and comply with data protection regulations.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Gimenez T, Sobral APT, Santos EM, Goncalves MLL, Ferri EP, Gallo JMAS, Horliana ACRT, Motta LJ, Imparato JCP, Bussadori SK. An investigator-blinded, 24-month, parallel-group, non-inferiority study to compare aesthetic restorations in primary anterior teeth in a paediatric dental clinic: study protocol for a randomised controlled trial. BMJ Open. 2025 Feb 6;15(2):e086200. doi: 10.1136/bmjopen-2024-086200. PMID 39915031